CLINICAL TRIAL: NCT05025046
Title: Prospective, Blinded, Multi-center Clincal Study of NGS-based Thyroscan Genomic Classifier in the Diagnosis of Thyroid Nodules
Brief Title: NGS-based Thyroscan Genomic Classifier in the Diagnosis of Thyroid Nodules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigen Biotech (Industry)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); Guangdong Provincial People's Hospital (Other); RenJi Hospital (Other); Zhejiang Provincial People's Hospital (Other); The First People's Hospital of Changzhou (Other); Shenzhen People's Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Sponsor
Other Study IDs: RigenBio
Record Dates: First submitted 2021-08-25; First posted 2021-08-27 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Thyroid Nodule; Thyroid Cancer
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultrasound findings of thyroid nodules classified as type 3 and 4a of TIRADS
  Interventions: Diagnostic Test: Thyroscan

INTERVENTIONS:
Diagnostic Test: Thyroscan — To evaluate the accuracy of Thyroscan in the differential diagnosis of benign and malignant thyroid nudules with abnormal ultrasound features.

SUMMARY:
The purpose of this study is to evaluate the accuracy of Thyroscan in the differential diagnosis of benign and malignant thyroid nodules with suspecious ultrasound features

DETAILED DESCRIPTION:
The prevalence of thyroid nodules by high-resolution ultrasound can be as high as 20%, though most of them are benign lesions, only about 5%~15% are malignant lesions. Based on 1.4 billion population in China, there are approximately 280 million thyroid nodule carriers, of which approximately 14~42 million are potential patients with thyroid cancer. Now thyroid cancer is the fastest growing cancer and the 4th most common cancer in women in China. Therefore, the key point in the evaluation of thyroid nodules is the differential diagnosis of benign and malignant nodules. At present, the commonly used imaging and cytological diagnostic techniques for thyroid nodules include ultrasound and ultrasound-guided fine needle aspiration biopsy (FNAB), as well as emerging molecular diagnostic techniques.

The purpose of this study is to evaluate the accuracy of Thyroscan in the diagnosis of benign and malignant thyroid nodules with suspecious ultrasound features. For patients who have signed an informed consent, the subjects undergo fine needle aspiration of thyroid nodules classified as C-TIRADS catagories 3 or 4a under the guidance of ultrasound or palpation before receiving surgical treatment. One needle is used to prepare cytological smear, and one needle is preserved and sent to Thyroscan detection. The histopathological is obtained as the "gold standerd" after surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients sign the informed consent form for participating in the reasearch study.
2. Patient's age is 18 years or older.
3. Ultrasound showed at least one thyroid nodule, and it was classified as C-TIRADS Category 3/4a.
4. The surgeon has evaluated the indications for surgery, and the subject is willing to receive surgical intervention in the medical institution.
5. Surgical indications include but are not limited to one of the following conditions: 1) Thyroid nodules are compressed or affect aesthetics; 2) The patient's subjective wishes require surgical removal of the nodules; 3) FNA samples with indeterminate cytology are classified as Bethesda III and IV, requiring diagnostic surgery; 4) After the investigator's assessment, there are other surgical indications.
6. Preoperative FNAB to obtain sufficient cells to meet FNA samples with indeterminate cytology are classified as Bethesda III and IV.
7. The final pathological diagnosis is obtained after surgury.

Exclusion Criteria:

1. The subject has a history of thyroid tumor.
2. The subject has swollen lymph nodes in the central area or/and lateral neck area.
3. The subject is not suitable for fine-needle aspiration biopsy and surgical treatment due to other conditions such as comorbid diseases.
4. FNAB interprets the thyroid nodule as Bethesda V and VI categories.
5. Subjects who intend to receive the radiofrequency ablation therapy.
6. Other conditions determined by the researcher that do not meet the criteria of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that ultrasound scan identified at least one thyroid nodule, which was classified as category 3 and 4a according to the C-TIRADS guideline.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
To evaluation of Thyroscan's performance in diagnosing thyroid nodules | June,2022
  To explore the sensitivity, specificity, positive predictive value, negative predictive value, consistency and Kappa value of Thyroscan in the diagnosis of thyroid nodules with ultrasound features classified as C-TIRADS category 3/4a.

SECONDARY OUTCOMES:
To compared with cytopathology and Thyroscan in diagnosing thyroid nodules. | June,2022
To explore the inter-observer heterogeneity when reviewing fine needle aspiration biopsy(FNAB) by two senior cytopathologists. | June,2022

OTHER OUTCOMES:
To explore the cost-effectiveness analysis of Thyroscan. | June,2022
To reveals the correlation between molecular landscape and clinical-pathological characteristics of thyroid nodules. | June,2022

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - The First Peple's Hospital of Changzhou, Changzhou, Jiangsu
  - Guangdong Provincial People's Hospital, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Shanghai Jiaotong University School of Medicine, Shanghai
  - Shenzhen People's Hospital, Shenzhen
  - Tianjin Medical University Center Hospital, Tianjin